CLINICAL TRIAL: NCT01378442
Title: The Relationship of Bone Strength and Fitness Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 95-1164B
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2011-05

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; bone density; bone strength
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high level training group (Experimental): receive high frequency fitness training program(Frequency: three times a week, Duration: 40 minutes).
  Interventions: Other: fitness training program
- low level training group (Experimental): will receive low frequency fitness training program(Frequency: 1-2 times a week, Duration: 40 minutes).
  Interventions: Other: fitness training program
- control (No Intervention): No intervention, but maintain usual physical activities

INTERVENTIONS:
Other: fitness training program — Experimental: high level training group. The experimental group received training for 40 min per day 3 times a week for 12 weeks. The hVCT program consisted of a 5-min warm-up exercise, twenty repetitions of sitting-to-standing movements, cycling for 20 min, and a cool-down exercise for 5 min.
  Experimental: low level training group. The experimental group received training for 40 min per day 1-2 times a week for 12 weeks. The program consisted of a 5-min warm-up exercise, twenty repetitions of sitting-to-standing movements, fitness training for 20 min, and a cool-down exercise for 5 min.
  Control:The control group will not receive fitness training program but maintain the usual life style.
  Arms: high level training group; low level training group

SUMMARY:
In the first year, all subjects received clinical assessments include subjective assessment, basic data, nutritional status and fitness assessments. Laboratory assessments include body composition, bone density(lumbar spine and femur by dual energy X-ray absorptiometry ), bone strength (by calcaneal ultrasound) and bone metabolism.

In the 2nd year, were randomized into three groups. The high level training group (20 children) will receive high frequency fitness training program(Frequency: three times one week, Duration: thirty minutes). The low level training group (20 children) will receive low frequency fitness training program(Frequency: two times one week, Duration: thirty minutes).The control group (20 children) will not receive fitness training program but maintain the usual life style.

In the 3rd year, all subjects received post-training clinical assessments include subjective assessment, basic data, nutritional status and fitness assessments. Laboratory assessments include body composition, bone density(lumbar spine and femur by dual energy X-ray absorptiometry ), bone strength (by calcaneal ultrasound) and bone metabolism.

These data provided in this study could establish the bone quality and fitness data of children with diplegic CP, and provide us to plan treatment strategies in the management of bone and fitness problems in the future.

DETAILED DESCRIPTION:
Malnutrition and motor impairment are common in children with cerebral palsy. Poor nutrition and motor impairment may further contribute to fitness impairment, low bone mineralization density (BMD), low bone strength, and even fractures in children with CP. To management of bone problems is based on the understanding the pathophysiology of bone mineralization or bone strength in CP.

Multiple factors, including nutritional factors (eg. nutritional status, body composition) and non-nutritional factors (eg. fitness, immobility, use of anticonvulsants) that may potentially have an impact on bone density/strength in children with CP However, there were few studies to investigate the relationship of bone strength and fitness in children with cerebral palsy in Taiwan. We hypothesized that fitness training may potentially have an impact on bone density/strength in children with CP. The purpose of this study is to further find out the relationship of bone quality and fitness training in children with CP.

We will collect 60 children with diplegic CP. The inclusion criteria include good cognition to comprehend the command and cooperation during examination and fitness training. The exclusion criteria were following as chromosomal abnormalities, active medical conditions such as pneumonia or others, poor tolerance during assessment and fitness training.

In the first year, all subjects received clinical assessments include subjective assessment, basic data, nutritional status and fitness assessments. Laboratory assessments include body composition, bone density(lumbar spine and femur by dual energy X-ray absorptiometry ), bone strength (by calcaneal ultrasound) and bone metabolism.

In the 2nd year, were randomized into three groups. The high level training group (20 children) will receive high frequency fitness training program(Frequency:three times one week, Duration: 40 minutes).The low level training group (20 children) will receive low frequency fitness training program(Frequency: 1-2 times one week, Duration: 40 minutes). The control group (20 children) will not receive fitness training program but maintain the usual life style.

In the 3rd year, all subjects received post-training clinical assessments include subjective assessment, basic data, nutritional status and fitness assessments. Laboratory assessments include body composition, bone density(lumbar spine and femur by dual energy X-ray absorptiometry ), bone strength (by calcaneal ultrasound) and bone metabolism.

These data provided in this study could establish the bone quality and fitness data of children with diplegic CP, and provide us to plan treatment strategies in the management of bone and fitness problems in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-18 years
* Good cognition to comprehend the command
* Good cooperation during examination and fitness training

Exclusion Criteria:

* children with recognized chromosomal abnormalities
* Active medical conditions such as pneumonia or others
* Poor tolerance during assessment and fitness training

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral Density Measurements | 12 and 24 weeks
  BMD in the lumbar spine and hip are measured with DXA. Standard scanning procedures were used for the lumbar spine. BMD measurements (g/cm2) were converted to age- and gender-normalized standard deviation scores (z scores).

SECONDARY OUTCOMES:
Children's Health Status | 12 and 24 weeks
  Children's Health Status Questionnaire
quality of life | 12 and 24 weeks
  Cerebral Palsy Quality of Life Questionnaire
Body composition | 12 and 24 weeks
  Body composition, lean body mass and body fat are measured
Muscle strength | 12 and 24 weeks
  Hand grasp assessment by the hand dynamometer Abdominal muscle strength by curling up
Flexibility | 12 and 24 weeks
  Forward bending distance during sitting position
Cardiopulmonary function | 12 and 24 weeks
  Measurement of times when performing stepping forward and backward for 1 minute. The changes of heart rate and blood pressure before and after stepping
Bone strength | 12 and 24 weeks
  Calcaneal bone strength BUA
Bone metabolism | 12 and 24 weeks
  Serum calcium, Phosphate,Serum intact parathyroid hormone (iPTH),Serum total alkaline phosphatase (ALP),Urine deoxypyridinoline(D-Pyr)
Motor function | 12 and 24 weeks
  BOTMP, GMFM
Muscle strength | 12 and 24 weeks
  isokinetic torque of knee flexor and extensor at different angular velocities

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, PhD, Principal Investigator — Department of Physical Medicine & Rehabilitation, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan